CLINICAL TRIAL: NCT02262520
Title: Effect of Apixaban on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: Phase 1 Drug Interaction Study of the Effect of Apixaban on the PK of Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-028
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: N/A - Healthy Subjects
MeSH Terms: interventions — apixaban; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: Digoxin (Experimental): Digoxin tablet by mouth on specified days
  Interventions: Drug: Digoxin
- Treatment B: Apixaban and Digoxin (Experimental): Apixaban and Digoxin tablets by mouth on specified days
  Interventions: Drug: Apixaban; Drug: Digoxin

INTERVENTIONS:
Drug: Apixaban
  Arms: Treatment B: Apixaban and Digoxin
Drug: Digoxin

SUMMARY:
The purpose of this study is to assess the effects of Apixaban on the Pharmacokinetics (PK) of multiple-dose Digoxin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

• Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECGs), and clinical laboratory determinations

Exclusion Criteria:

• Any significant acute or chronic medical illness, history of important arrhythmias, history or evidence of abnormal bleeding or coagulation disorders, significant head injury within the last 2 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Apixaban and Digoxin plasma concentration | Days 8-21
  Blood samples for Digoxin were collected on Days 8, 9, 10, 11, 18, 19, 20 & 21 Urine samples for Digoxin were collected for 24 hours post dose on Days 10 & 20. Blood samples for Apixaban concentration were collected on Days 18-20

SECONDARY OUTCOMES:
Safety and Tolerability based on medical review of adverse event reports and the results of vital sign measurements, physical examinations, electrocardiograms, digoxin concentrations,and clinical laboratory tests | Days 1-22

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb